CLINICAL TRIAL: NCT02219685
Title: A Phase 2, Single-Center, Double-Blind, Placebo-Controlled, Randomized Study to Investigate the Effect of Ledipasvir/Sofosbuvir Fixed-Dose Combination on Cerebral Metabolism and Neurocognition in Treatment-Naive and Treatment-Experienced Subjects With Chronic Genotype 1 HCV Infection
Brief Title: Ledipasvir/Sofosbuvir Fixed-Dose Combination on Cerebral Metabolism and Neurocognition in Treatment-Naive and Treatment-Experienced Participants With Chronic Genotype 1 HCV Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GS-US-337-1445
Record Dates: First submitted 2014-08-15; First posted 2014-08-19 (Estimated); Results first posted 2016-11-30 (Estimated); Last update posted 2018-11-16 (Actual); Status verified 2016-10

CONDITIONS: Hepatitis C Virus Infection
MeSH Terms: conditions — Hepatitis C | interventions — ledipasvir, sofosbuvir drug combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- LDV/SOF (Experimental): Participants will receive LDV/SOF FDC for 12 weeks.
  Interventions: Drug: LDV/SOF
- Placebo (Placebo Comparator): Participants will receive LDV/SOF placebo for 12 weeks.
  Interventions: Drug: Placebo
- Open-Label Treatment Phase (Experimental): Following Posttreatment Week 4, participants in the placebo group will be offered open-label treatment with LDV/SOF FDC for 12 weeks.
  Interventions: Drug: LDV/SOF

INTERVENTIONS:
Drug: LDV/SOF — 90/400 mg FDC tablet administered orally once daily
  Other Names: Harvoni®; GS-5885/GS-7977
  Arms: LDV/SOF; Open-Label Treatment Phase
Drug: Placebo — Tablet administered orally once daily
  Arms: Placebo

SUMMARY:
The primary objectives of this study are to evaluate the effect of sustained virologic response (SVR) on cerebral metabolism as determined by magnetic resonance spectroscopy (MRS) and on neurocognition as measured by neurocognitive tests. This study will also evaluate the antiviral efficacy, safety, and tolerability of ledipasvir/sofosbuvir (LDV/SOF) fixed-dose combination (FDC) for 12 weeks in treatment-naive or treatment-experienced adults.

During the blinded treatment phase, participants will be randomized 2:1 to receive LDV/SOF FDC or placebo for 12 weeks. After the unblinding at the Posttreatment Week 4 visit, participants in the placebo group will be offered open-label treatment of LDV/SOF FDC for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Chronic HCV infection (≥ 6 months) documented by prior medical history or liver biopsy
* Chronic genotype 1 HCV infection
* Screening laboratory values within defined thresholds
* Use of protocol-specified method(s) of contraception if female of childbearing potential or sexually active male

Exclusion Criteria:

* Clinically-significant illness (other than HCV) or any other major medical disorder that may interfere with treatment, assessment, or compliance with the protocol. Current or prior history of any of the following:

  * Hepatic decompensation
  * Solid organ transplantation
  * Significant pulmonary or cardiac disease
  * Chronic liver disease of a non-HCV etiology
  * Hepatocellular carcinoma (HCC)
  * Infection with hepatitis B virus (HBV)
  * Infection with human immunodeficiency virus (HIV)
  * History of recent epilepsy (within 2 years of screening) or cerebral vascular accident (CVA)
  * Structural brain damage
* Presence of cirrhosis
* Contraindication to MRI
* Pregnant or nursing female
* Prior treatment NS5A directly-acting antiviral agent. Any interferon (IFN)-containing regimen within 8 weeks of Screening

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2014-08; Primary Completion 2015-08 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benedetta Massetto, MD, Study Director — Gilead Sciences
Locations (1):
- Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at http://www.gilead.com/research/disclosure-and-transparency.
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: http://www.gilead.com/research/disclosure-and-transparency

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 1 study site in the United States. The first participant was screened on 25 August 2014. The last study visit occurred on 07 April 2016.
Pre-assignment Details: 54 participants were screened.
Groups:
- LDV/SOF: Ledipasvir/sofosbuvir (LDV/SOF) (90/400 mg) fixed-dose combination (FDC) tablet once daily for 12 weeks
- Placebo, Followed by Open-Label LDV/SOF: LDV/SOF placebo tablet once daily for 12 weeks, followed by LDV/SOF (90/400 mg) FDC tablet once daily for 12 weeks
Period: Blinded Treatment Phase
Arm/Group | LDV/SOF | Placebo, Followed by Open-Label LDV/SOF
Started | 26 | 14
Completed | 24 | 14
Not Completed | 2 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrew Consent | 1 | 0
Period: Open-Label (After Posttreatment Week 4)
Arm/Group | LDV/SOF | Placebo, Followed by Open-Label LDV/SOF
Started | 0 (Only participants from the Placebo arm were eligible to enroll in the Open-Label Phase.) | 14
Completed | 0 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: participants who were randomized into the study and received at least 1 dose of study drug.
Groups:
- LDV/SOF: LDV/SOF (90/400 mg) FDC tablet once daily for 12 weeks
- Placebo: LDV/SOF placebo tablet once daily for 12 weeks, followed by LDV/SOF (90/400 mg) FDC tablet once daily for 12 weeks
- Total: Total of all reporting groups
Arm/Group | LDV/SOF | Placebo | Total
Number analyzed (Participants) | 26 | 14 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 44 (12.4) | 47 (9.8) | 45 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 9 | 21
  Male | 14 | 5 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 3
  Not Hispanic or Latino | 23 | 14 | 37
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Black or African American | 3 | 1 | 4
  White | 23 | 13 | 36
Prior HCV Treatment Experience [Number; unit: participants]
  Treatment-Naive | 15 | 8 | 23
  Treatment-Experienced | 11 | 6 | 17
HCV Genotype [Number; unit: participants]
  Genotype 1a | 23 | 12 | 35
  Genotype 1b | 3 | 2 | 5
IL28B Status [Number; unit: participants] — The CC, CT, and TT alleles are different forms of the IL28b gene.
  participants
    CC | 4 | 3 | 7
    CT | 19 | 8 | 27
    TT | 3 | 3 | 6
HCV RNA [Mean (Standard Deviation); unit: log10 IU/mL] | 6.2 (0.57) | 6.4 (0.62) | 6.3 (0.58)
HCV RNA Category [Number; unit: participants]
  < 800,000 IU/mL | 9 | 3 | 12
  ≥ 800,000 IU/mL | 17 | 11 | 28

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Magnetic Resonance Spectroscopy (MRS) Metabolic Ratio at 4 Weeks After Discontinuation of Therapy: NAA + NAAG
Description: MRS was analyzed in the LCmodel program and measured in 3 specific areas of brain (basal ganglia, frontal cortex, and dorsolateral prefrontal cortex). The cerebral metabolic signal N-acetylaspartate (NAA) + N-acetylaspartylglutamate (NAAG) was analyzed. Spectroscopy results are expressed as metabolic ratio with creatine used as the control metabolite, so there are no units of measure.
Time Frame: Baseline; Posttreatment Week 4
Population: Full Analysis Set: participants who were randomized into the study and received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: ratio
Groups:
- Blinded Phase: LDV/SOF: LDV/SOF (90/400 mg) FDC tablet once daily for 12 weeks during the Blinded Treatment Phase
- Blinded Phase: Placebo: LDV/SOF placebo tablet once daily for 12 weeks during the Blinded Treatment Phase
Arm/Group | Blinded Phase: LDV/SOF | Blinded Phase: Placebo
Number analyzed (Participants) | 26 | 14
ratio
  Basal Ganglia | -0.03 (0.085) | -0.01 (0.147)
  Frontal Cortex | -0.03 (0.201) | -0.09 (0.279)
  Dorsolateral Prefrontal Cortex | 0.00 (0.154) | -0.01 (0.142)
Statistical Analysis 1: Comparison: Blinded Phase: LDV/SOF vs Blinded Phase: Placebo; Test type: Superiority or Other; p = 0.58, t-test, 2 sided — This p-value for treatment effect on basal ganglia was based on a two sample t-test assuming equal variances
Statistical Analysis 2: Comparison: Blinded Phase: LDV/SOF vs Blinded Phase: Placebo; Test type: Superiority or Other; p = 0.48, t-test, 2 sided — This p-value for treatment effect on frontal cortex was based on a two sample t-test assuming equal variances
Statistical Analysis 3: Comparison: Blinded Phase: LDV/SOF vs Blinded Phase: Placebo; Test type: Superiority or Other; p = 0.96, t-test, 2 sided — This p-value for treatment effect on dorsolateral prefrontal cortex was based on a two sample t-test assuming equal variances

2. Primary Outcome: Change From Baseline in MRS Metabolic Ratio at 4 Weeks After Discontinuation of Therapy: Choline
Description: MRS was analyzed in the LCmodel program and measured in 3 specific areas of brain (basal ganglia, frontal cortex, and dorsolateral prefrontal cortex). The cerebral metabolic signal choline was analyzed. Spectroscopy results are expressed as metabolic ratio with creatine used as the control metabolite, so there are no units of measure.
Time Frame: Baseline; Posttreatment Week 4
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Blinded Phase: LDV/SOF | Blinded Phase: Placebo
Number analyzed (Participants) | 26 | 14
ratio
  Basal Ganglia | -0.01 (0.020) | 0.00 (0.029)
  Frontal Cortex | 0.01 (0.033) | 0.00 (0.055)
  Dorsolateral Prefrontal Cortex | 0.00 (0.029) | 0.01 (0.023)
Statistical Analysis 1: Comparison: Blinded Phase: LDV/SOF vs Blinded Phase: Placebo; Test type: Superiority or Other; p = 0.54, t-test, 2 sided — This p-value for treatment effect on basal ganglia was based on a two sample t-test assuming equal variances
Statistical Analysis 2: Comparison: Blinded Phase: LDV/SOF vs Blinded Phase: Placebo; Test type: Superiority or Other; p = 0.57, t-test, 2 sided — This p-value for treatment effect on frontal cortex was based on a two sample t-test assuming equal variances
Statistical Analysis 3: Comparison: Blinded Phase: LDV/SOF vs Blinded Phase: Placebo; Test type: Superiority or Other; p = 0.63, t-test, 2 sided — [p-value comment as in outcome 1, analysis 3]

3. Primary Outcome: Change From Baseline in MRS Metabolic Ratio at 4 Weeks After Discontinuation of Therapy: Myoinositol
Description: MRS was analyzed in the LCmodel program and measured in 3 specific areas of brain (basal ganglia, frontal cortex, and dorsolateral prefrontal cortex). The cerebral metabolic signal myoinositol was analyzed. Spectroscopy results are expressed as metabolic ratio with creatine used as the control metabolite, so there are no units of measure.
Time Frame: Baseline; Posttreatment Week 4
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Blinded Phase: LDV/SOF | Blinded Phase: Placebo
Number analyzed (Participants) | 26 | 14
ratio
  Basal Ganglia | 0.02 (0.110) | 0.00 (0.157)
  Frontal Cortex | -0.01 (0.207) | 0.08 (0.156)
  Dorsolateral Prefrontal Cortex | -0.02 (0.112) | 0.00 (0.104)
Statistical Analysis 1: Comparison: Blinded Phase: LDV/SOF vs Blinded Phase: Placebo; Test type: Superiority or Other; p = 0.70, t-test, 2 sided — This p-value for treatment effect on basal ganglia was based on a two sample t-test assuming equal variances
Statistical Analysis 2: Comparison: Blinded Phase: LDV/SOF vs Blinded Phase: Placebo; Test type: Superiority or Other; p = 0.21, t-test, 2 sided — This p-value for treatment effect on frontal cortex was based on a two sample t-test assuming equal variances
Statistical Analysis 3: Comparison: Blinded Phase: LDV/SOF vs Blinded Phase: Placebo; Test type: Superiority or Other; p = 0.59, t-test, 2 sided — [p-value comment as in outcome 1, analysis 3]

4. Primary Outcome: Change From Baseline in Neurocognitive Function at 4 Weeks After Discontinuation of Therapy: Memory T Score
Description: Neurocognitive function tests were administered by a licensed clinician. The sum of following neurocognitive test scores was used to determine the Memory T Score: visuospatial memory immediate total T score (BVMTTTs), visuospatial memory delayed T score (BVMTTDTS), verbal memory total T score (HVLTTTS), and verbal memory delayed T score (HVLTDTS).
  For this analysis, Memory T Score (total) ranged from 80 to 320, with higher scores indicating better memory.
Time Frame: Baseline; Posttreatment Week 4
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Blinded Phase: LDV/SOF | Blinded Phase: Placebo
Number analyzed (Participants) | 26 | 14
units on a scale | -3.88 (19.15) | 7.93 (23.63)
Statistical Analysis 1: Comparison: Blinded Phase: LDV/SOF vs Blinded Phase: Placebo; Test type: Superiority or Other; p = 0.0795, ANCOVA — The p-value was from ANCOVA model for change from baseline with treatment group and baseline as covariates

5. Primary Outcome: Change From Baseline in Neurocognitive Function at 4 Weeks After Discontinuation of Therapy: Attention Scaled Score
Description: Neurocognitive function tests were administered by a licensed clinician. The sum of following neurocognitive test scores was used to determine the Attention Scaled Score: forward digit span scaled score (FSCORESS), backward digit span scaled score (BSCORESS), and symbol span total scaled score (SYMSPSS).
  For this analysis, Attention Scaled Score (total) ranged from 3 to 57, with higher scores indicating better working memory capacity and control.
Time Frame: Baseline; Posttreatment Week 4
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Blinded Phase: LDV/SOF | Blinded Phase: Placebo
Number analyzed (Participants) | 26 | 14
units on a scale | 0.73 (4.29) | 1.43 (3.34)
Statistical Analysis 1: Comparison: Blinded Phase: LDV/SOF vs Blinded Phase: Placebo; Test type: Superiority or Other; p = 0.7007, ANCOVA — The p-value was from ANCOVA model for change from baseline with treatment group and baseline as covariates

6. Primary Outcome: Change From Baseline in Neurocognitive Function at 4 Weeks After Discontinuation of Therapy: Executive 1 Processing Speed
Description: Neurocognitive function tests were administered by a licensed clinician. The sum of following neurocognitive test scores was used to determine the Executive 1 Processing Speed score: symbol search total scaled score (SSSS) and trails A total raw score (TrailARS).
  For this analysis, Executive 1 Processing Speed score (total) ranged from 1 to 108, with lower scores indicating better executive control.
Time Frame: Baseline; Posttreatment Week 4
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Blinded Phase: LDV/SOF | Blinded Phase: Placebo
Number analyzed (Participants) | 26 | 14
units on a scale | 1.96 (5.71) | 4.00 (7.27)
Statistical Analysis 1: Comparison: Blinded Phase: LDV/SOF vs Blinded Phase: Placebo; Test type: Superiority or Other; p = 0.2677, ANCOVA — The p-value was ANCOVA model for change from baseline with treatment group and baseline as covariates

7. Primary Outcome: Change From Baseline in Neurocognitive Function at 4 Weeks After Discontinuation of Therapy: Executive 2 Conceptual Shift and Initiation
Description: Neurocognitive function tests were administered by a licensed clinician. The sum of following neurocognitive test scores was used to determine the Executive 2 Conceptual Shift and Initiation score: trails B raw score (TrailBRS), age & education adjusted raw score (FASadj), color word interference score (time) (CWTrial3), and color word interference/shifting score (time) (CWTrial4).
  For this analysis, Executive 2 Conceptual Shift and Initiation score (total) ranged from 1 to 570, with lower scores indicating better executive control.
Time Frame: Baseline; Posttreatment Week 4
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Blinded Phase: LDV/SOF | Blinded Phase: Placebo
Number analyzed (Participants) | 26 | 14
units on a scale | -13.04 (21.03) | -12.43 (15.38)
Statistical Analysis 1: Comparison: Blinded Phase: LDV/SOF vs Blinded Phase: Placebo; Test type: Superiority or Other; p = 0.9870, ANCOVA — The p-value was from ANCOVA model for change from baseline with treatment group and baseline as covariates

8. Primary Outcome: Change From Baseline in Neurocognitive Function at 4 Weeks After Discontinuation of Therapy: Motor
Description: Neurocognitive function tests were administered by a licensed clinician. The sum of following neurocognitive test scores was used to determine the Motor score: dominant hand fine motor speed (time) (DomHtot) and non-dominant hand fine motor speed (time) (nonDOMHtot).
  For this analysis, Motor score (total) ranged from 20 to 600, with lower scores indicating better fine motor speed.
Time Frame: Baseline; Posttreatment Week 4
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Blinded Phase: LDV/SOF | Blinded Phase: Placebo
Number analyzed (Participants) | 26 | 14
units on a scale | -10.00 (17.47) | -6.00 (17.16)
Statistical Analysis 1: Comparison: Blinded Phase: LDV/SOF vs Blinded Phase: Placebo; Test type: Superiority or Other; p = 0.3388, ANCOVA — The p-value was from ANCOVA model for change from baseline with treatment group and baseline as covariates

9. Secondary Outcome: Percentage of Participants With Sustained Virologic Response (SVR) at 4, 12, and 24 Weeks After Discontinuation of Therapy (SVR4, SVR12, and SVR24)
Description: SVR4, SVR12, and SVR24 were defined as HCV RNA < the lower limit of quantitation (LLOQ; ie, 15 IU/mL) at 4, 12, and 24 weeks after stopping study treatment with LDV/SOF, respectively.
Time Frame: Posttreatment Weeks 4, 12, and 24
Population: Full Analysis Set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Open-Label Phase: LDV/SOF: LDV/SOF (90/400 mg) FDC tablet once daily for 12 weeks during the Open-Label Treatment Phase
Arm/Group | Blinded Phase: LDV/SOF | Open-Label Phase: LDV/SOF
Number analyzed (Participants) | 26 | 14
percentage of participants
  SVR4 | 96.2 [80.4 to 99.9] | 100.0 [76.8 to 100.0]
  SVR12 | 92.3 [74.9 to 99.1] | 100.0 [76.8 to 100.0]
  SVR24 | 92.3 [74.9 to 99.1] | 100.0 [76.8 to 100.0]

10. Secondary Outcome: Change From Baseline in Neurocognitive Function at 24 Weeks After Discontinuation of Therapy: Memory T Score
Description: as for outcome 4
Time Frame: Baseline; Posttreatment Week 24
Population: Participants in the Full Analysis Set with available data were analyzed. Data for the "Open-Label Phase: LDV/SOF" group are not presented because this group did not have a Posttreatment Week 24 visit after receiving placebo. These participants were enrolled into the Open-Label Phase after Posttreatment Week 4.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Blinded Phase: LDV/SOF
Number analyzed (Participants) | 24
units on a scale | -17.42 (31.57)

11. Secondary Outcome: Change From Baseline in Neurocognitive Function at 24 Weeks After Discontinuation of Therapy: Attention Scaled Score
Description: as for outcome 5
Time Frame: Baseline; Posttreatment Week 24
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Blinded Phase: LDV/SOF
Number analyzed (Participants) | 24
units on a scale | 1.42 (0.36)

12. Secondary Outcome: Change From Baseline in Neurocognitive Function at 24 Weeks After Discontinuation of Therapy: Executive 1 Processing Speed
Description: as for outcome 6
Time Frame: Baseline; Posttreatment Week 24
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Blinded Phase: LDV/SOF
Number analyzed (Participants) | 24
units on a scale | 4.00 (7.95)

13. Secondary Outcome: Change From Baseline in Neurocognitive Function at 24 Weeks After Discontinuation of Therapy: Executive 2 Conceptual Shift and Initiation
Description: as for outcome 7
Time Frame: Baseline; Posttreatment Week 24
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Blinded Phase: LDV/SOF
Number analyzed (Participants) | 24
units on a scale | -16.67 (35.12)

14. Secondary Outcome: Change From Baseline in Neurocognitive Function at 24 Weeks After Discontinuation of Therapy: Motor
Description: as for outcome 8
Time Frame: Baseline; Posttreatment Week 24
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Blinded Phase: LDV/SOF
Number analyzed (Participants) | 24
units on a scale | -9.21 (17.74)

15. Secondary Outcome: Change From Baseline in Health-Related Quality of Life at 4 and 24 Weeks After Discontinuation of Therapy as Assessed by Short Form 36 (SF-36) Health Survey Scale - Physical Component Score
Description: The SF-36 Health Survey is a self-reporting, multi-item scale measuring 8 health concepts: 1) physical functioning, 2) role limitations due to physical health problems, 3) bodily pain, 4) general health, 5) vitality (energy/fatigue), 6) social functioning, 7) role limitations due to emotional problems and 8) mental health (psychological distress and psychological well-being). The first 6 concepts constitute the physical component summary. The total score is an average of the individual question scores, which are scaled 0-100 with lower scores representing more disability and higher scores representing less disability.
Time Frame: Baseline; Posttreatment Weeks 4 and 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Blinded Phase: LDV/SOF | Blinded Phase: Placebo
Number analyzed (Participants) | 26 | 14
units on a scale
  Baseline (LDV/SOF: N =25; Placebo: N =14) | 53.8 (5.51) | 56.2 (4.42)
  Change at PT Wk 4 (LDV/SOF: N =25; Placebo: N =14) | 1.1 (3.73) | -0.1 (4.48)
  Change at PT Wk 24 (LDV/SOF: N =23; Placebo: NA) | 1.5 (4.13) | NA (NA) — Participants in the Placebo group did not have a Posttreatment Week 24 visit because they were enrolled into the Open-Label Phase after Posttreatment Week 4.

16. Secondary Outcome: Change From Baseline in Health-Related Quality of Life at 4 and 24 Weeks After Discontinuation of Therapy as Assessed by SF-36 Health Survey Scale - Mental Component Score
Description: The SF-36 Health Survey is a self-reporting, multi-item scale measuring 8 health concepts: 1) physical functioning, 2) role limitations due to physical health problems, 3) bodily pain, 4) general health, 5) vitality (energy/fatigue), 6) social functioning, 7) role limitations due to emotional problems and 8) mental health (psychological distress and psychological well-being). The last 5 concepts constitute the mental component summary. The total score is an average of the individual question scores, which are scaled 0-100 with lower score representing more disability and higher scores representing less disability.
Time Frame: Baseline; Posttreatment (PT) Weeks 4 and 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Blinded Phase: LDV/SOF | Blinded Phase: Placebo
Number analyzed (Participants) | 26 | 14
units on a scale
  Baseline (LDV/SOF: N = 25; Placebo: N = 14) | 52.5 (6.25) | 50.9 (10.26)
  Change at PT Wk 4 (LDV/SOF: N =25; Placebo: N =14) | 1.9 (4.86) | -2.9 (9.31)
  Change at PT Wk 24 (LDV/SOF: N =23; Placebo: NA) | 4.7 (5.77) | NA (NA) — Participants in the Placebo group did not have a Posttreatment Week 24 visit because they were enrolled into the Open-Label Phase after Posttreatment Week 4.

17. Secondary Outcome: Change From Baseline in Health-Related Quality of Life at 4 and 24 Weeks After Discontinuation of Therapy as Assessed by Chronic Liver Disease Questionnaire - HCV (CLDQ-HCV)
Description: The CLDQ-HCV is a disease-specific questionnaire measuring health-related quality of life. CLDQ-HCV scores are calculated using participant responses to 29 questions divided into 4 domains: Activity/Energy, Emotion, Worry, and Systemic. An overall CLDQ-HCV score is calculated by taking the mean of all domain scores. Overall CLDQ-HCV scores range between 1 and 7, with higher scores representing better quality of life.
Time Frame: Baseline; Posttreatment Weeks 4 and 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Blinded Phase: LDV/SOF | Blinded Phase: Placebo
Number analyzed (Participants) | 26 | 14
units on a scale
  Baseline (LVD/SOF: N =26; Placebo: N =14) | 5.8 (0.89) | 6.0 (0.78)
  Change at PT Wk 4 (LVD/SOF: N =26; Placebo: N =14) | 0.4 (0.61) | -0.1 (0.50)
  Change at PT Wk 24 (LVD/SOF: N =24; Placebo: NA) | 0.7 (0.77) | NA (NA) — Participants in the Placebo group did not have a Posttreatment Week 24 visit because they were enrolled into the Open-Label Phase after Posttreatment Week 4.

18. Secondary Outcome: Change From Baseline in Health-Related Quality of Life at 4 and 24 Weeks After Discontinuation of Therapy as Assessed by Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-F)
Description: The FACIT-Fatigue score was measured using a 40-item questionnaire that assesses self-reported fatigue and its impact upon daily activities and function. Participants scored each item on a 5-point scale from 0 (Not at all) to 4 (Very much). The FACIT-F total score was calculated by taking the sum of all 40 individual scores and ranged from 0-160, with higher scores indicating better quality of life.
Time Frame: Baseline; Posttreatment Weeks 4 and 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Blinded Phase: LDV/SOF | Blinded Phase: Placebo
Number analyzed (Participants) | 26 | 14
units on a scale
  Baseline (LDV/SOF: N =26; Placebo: N =14) | 94.7 (12.12) | 97.0 (8.72)
  Change at PT Wk 4 (LDV/SOF: N =26; Placebo: N =14) | 3.1 (8.43) | -4.4 (9.87)
  Change at PT Wk 24 (LDV/SOF: N =24; Placebo: NA) | 5.9 (9.04) | NA (NA) — Participants in the Placebo group did not have a Posttreatment Week 24 visit because they were enrolled into the Open-Label Phase after Posttreatment Week 4.

19. Secondary Outcome: Change From Baseline in Health-Related Quality of Life at 4 and 24 Weeks After Discontinuation of Therapy as Assessed by Work Productivity and Activity Impairment Questionnaire, Hepatitis C (WPAI: Hepatitis C) - Overall Work Impairment
Description: Impairment in overall work productivity was measured using the WPAI: Hepatitis C questionnaire completed by participants during study visits throughout the study. This questionnaire measured the effect of hepatitis C on the ability to work and perform regular activities. Overall work impairment is expressed as a percentage and ranges from 0% (no effect) to 100% (completely prevented from working).
Time Frame: Baseline; Posttreatment Weeks 4 and 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Blinded Phase: LDV/SOF | Blinded Phase: Placebo
Number analyzed (Participants) | 26 | 14
units on a scale
  Baseline (LDV/SOF: N =24; Placebo: N =10) | 12.6 (28.16) | 4.0 (9.66)
  Change at PT Wk 4 (LDV/SOF: N =21; Placebo: N =10) | -11.5 (27.31) | 13.0 (22.63)
  Change at PT Wk 24 (LDV/SOF: N =20; Placebo: NA) | -3.6 (34.01) | NA (NA) — Participants in the Placebo group did not have a Posttreatment Week 24 visit because they were enrolled into the Open-Label Phase after Posttreatment Week 4.

20. Secondary Outcome: Change From Baseline in Health-Related Quality of Life at 4 and 24 Weeks After Discontinuation of Therapy as Assessed by WPAI: Hepatitis C - Activity Impairment
Description: Activity impairment was measured using the WPAI: Hepatitis C questionnaire completed by participants during study visits throughout the study. This questionnaire measured the effect of hepatitis C on the ability to work and perform regular activities. Overall activity impairment is expressed as a percentage and ranges from 0% (no effect) to 100% (completely prevented from performing regular activities).
Time Frame: Baseline; Posttreatment Weeks 4 and 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Blinded Phase: LDV/SOF | Blinded Phase: Placebo
Number analyzed (Participants) | 26 | 14
units on a scale
  Baseline (LDV/SOF: N =26; Placebo: N =13) | 10.0 (24.17) | 2.3 (8.32)
  Change at PT Wk 4 (LDV/SOF: N =26; Placebo: N =13) | -6.9 (23.28) | 6.9 (11.82)
  Change at PT Wk 24 (LDV/SOF: N =20; Placebo: NA) | -6.1 (19.48) | NA (NA) — Participants in the Placebo group did not have a Posttreatment Week 24 visit because they were enrolled into the Open-Label Phase after Posttreatment Week 4.

21. Secondary Outcome: Change From Pre-treatment Assessment in Mood Related Assessment at 4 and 24 Weeks After Discontinuation of Therapy as Assessed by Beck Depression Inventory-II (BDI-II)
Description: The BDI-II is a 21-item self-report instrument for measuring the severity of depression. Each item is rated on a 4-point scale ranging from 0 to 3. The item scores are summed to yield a derived total score that can range from 0 to 63 with lower values indicating less depression.
Time Frame: Baseline; Posttreatment Weeks 4 and 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Blinded Phase: LDV/SOF | Blinded Phase: Placebo
Number analyzed (Participants) | 25 | 14
units on a scale
  Baseline | 4.20 (4.73) | 4.29 (5.98)
  Change at Posttreatment Week 4 | -2.40 (3.77) | 0.29 (5.04)
  Change at Posttreatment Week 24 | -2.74 (3.95) | NA (NA) — Participants in the Placebo group did not have a Posttreatment Week 24 visit because they were enrolled into the Open-Label Phase after Posttreatment Week 4.

22. Secondary Outcome: Change From Pre-treatment Assessment in Mood Related Assessment at 4 and 24 Weeks After Discontinuation of Therapy as Assessed by Beck Hopelessness Scale (BHS)
Description: The BHS is a 20-item scale for measuring the extent of negative attitudes about the future (pessimism) as perceived by adolescents and adults. The BHS consists of 20 true-false statements. Each of the 20 statements is scored 1 or 0. Of the 20 true-false statements, 9 are keyed FALSE, and 11 are keyed TRUE to indicate endorsement of pessimism about the future. The item scores are summed to yield a total score that can range from 0 to 20 with higher scores indicating greater hopelessness.
Time Frame: Baseline; Posttreatment Weeks 4 and 24
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Blinded Phase: LDV/SOF | Blinded Phase: Placebo
Number analyzed (Participants) | 26 | 14
units on a scale
  Baseline | 1.27 (1.40) | 1.36 (1.55)
  Change at Posttreatment Week 4 | -0.04 (1.43) | 0.14 (1.56)
  Change at Posttreatment Week 24 | -0.04 (0.91) | NA (NA) — Participants in the Placebo group did not have a Posttreatment Week 24 visit because they were enrolled into the Open-Label Phase after Posttreatment Week 4.

ADVERSE EVENTS:
Time Frame: Blinded Treatment Phase: Up to 12 weeks plus 30 days; Open-Label Treatment Phase: Up to 12 weeks plus 30 days
Description: Safety Analysis Set
Groups:
- LDV/SOF (Blinded Phase): LDV/SOF (90/400 mg) FDC tablet once daily for 12 weeks
- Placebo (Blinded Phase): LDV/SOF placebo tablet once daily for 12 weeks
- LDV/SOF (Open-Label Phase), Following Placebo in Blinded Phase: LDV/SOF (90/400 mg) FDC tablet once daily for 12 weeks during the Open-Label Treatment Phase
Arm/Group | LDV/SOF (Blinded Phase) | Placebo (Blinded Phase) | LDV/SOF (Open-Label Phase), Following Placebo in Blinded Phase
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 20/26 | 12/14 | 9/14
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LDV/SOF (Blinded Phase) (N=26) | Placebo (Blinded Phase) (N=14) | LDV/SOF (Open-Label Phase), Following Placebo in Blinded Phase (N=14)
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 2 | 3
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1
Faeces pale (Gastrointestinal disorders) | 0 | 1 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 5 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 0
Chills (General disorders) | 0 | 1 | 0
Fatigue (General disorders) | 5 | 6 | 1
Laryngitis (Infections and infestations) | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 6 | 3 | 2
Respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Blood pressure increased (Investigations) | 2 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 0 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Disturbance in attention (Nervous system disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 2 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 5 | 2 | 3
Restless legs syndrome (Nervous system disorders) | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 2 | 1
Irritability (Psychiatric disorders) | 0 | 1 | 0
Orchitis noninfective (Reproductive system and breast disorders) | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Tooth extraction (Surgical and medical procedures) | 0 | 1 | 0
Hypertension (Vascular disorders) | 2 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years